CLINICAL TRIAL: NCT01713205
Title: Identifying Severe Trauma Patients at High Risk of Post-traumatic Complications
Brief Title: Prediction Study of Complications After Severe Trauma
Acronym: PSCAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jiang Jianxin (Other)
Collaborators: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); Chongqing Emergency Medical Center (Other); Huazhong University of Science and Technology (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Kunming general Hospital of Chengdu Military Region (Unknown); The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Jiang Jianxin, Principal Investigator, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Organization: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Other Study IDs: Jiang-2012BAI11B01; 2012BAI11B01 (Other Grant/Funding Number: Five-twelfth National Science and Technology Support Program)
Record Dates: First submitted 2012-10-18; First posted 2012-10-24 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Trauma; Sepsis; Multiple Organ Dysfunction Syndrome
Keywords: trauma ; sepsis; Multiple Organ Dysfunction Syndrome; Prediction; risk
MeSH Terms: conditions — Wounds and Injuries; Sepsis; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, urine and tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate a clinically and economically most effective diagnostic algorithm for prediction of post-traumatic complications in a multicenter sample of severe trauma patients.

DETAILED DESCRIPTION:
Trauma is a major public health problem worldwide, ranking as the fourth leading cause of death. One of the most serious complications of major trauma is sepsis, which often induces sequential multiple organ dysfunction syndrome (MODS). There were still no specific biomarkers to predict the susceptibility of complications and outcomes, which leading to the limited prevention methods and the high mortality rate of severe trauma patients. Previous studies from our and other group have found some sepsis and MODS predictors, including genetic polymorphisms, serum cytokines and cell-surface markers. The purposes of this multi-center observational study is to select biomarkers and evaluate a clinically and economically most effective diagnostic algorithm for prediction of complications in severe trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* age> 16 years old and <65 years old
* severe trauma patients (AIS ≧3 or ISS≧16)
* admission within 48 hours after injury
* given and signed informed consent

Exclusion Criteria:

* died within 48h after injury
* being pregnant or lactating
* chronic organ dysfunction comorbidities
* long-term anticoagulant therapy before injury
* presence of immunosuppression before injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult severe trauma patients with no serious co-morbidity
Sampling Method: Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2012-10; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
morbidity rate of complications after trauma (including sepsis and MODS) | patients will be followed for the duration of hospital stay, an expected average of 3 weeks

SECONDARY OUTCOMES:
survival | witnin 30 days and 60 days after injury

CONTACTS AND LOCATIONS:
Overall Officials: Jianxin Jiang, MD,PhD, Principal Investigator — Daping Hospital/Research Institute of Surgery, Third Military Medical University
Locations (6):
- China (6):
  - Department of Emergency Surgery, The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei
  - Kunming General Hospital of Chengdu Military Region, Kunming, Yunnan
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Chongqing Emergency Medical Center, Chongqing
  - Daping Hospital / Research Institute of Surgery, the Third Military Medical University, Chongqing

REFERENCES:
- [Background] Gu W, Jiang J. Genetic polymorphisms and posttraumatic complications. Comp Funct Genomics. 2010;2010:814086. doi: 10.1155/2010/814086. Epub 2011 Jan 11. PMID 21274447
- [Result] Gu W, Zeng L, Zhang LY, Jiang DP, Du DY, Hu P, Wang HY, Liu Q, Huang SN, Jiang JX. Association of interleukin 4 -589T/C polymorphism with T(H)1 and T(H)2 bias and sepsis in Chinese major trauma patients. J Trauma. 2011 Dec;71(6):1583-7. doi: 10.1097/TA.0b013e3182115034. PMID 21460743
- [Result] Chen KH, Zeng L, Gu W, Zhou J, Du DY, Jiang JX. Polymorphisms in the toll-like receptor 9 gene associated with sepsis and multiple organ dysfunction after major blunt trauma. Br J Surg. 2011 Sep;98(9):1252-9. doi: 10.1002/bjs.7532. Epub 2011 Jun 1. PMID 21633947
- [Result] Zeng L, Zhang AQ, Gu W, Chen KH, Jiang DP, Zhang LY, Du DY, Hu P, Huang SN, Wang HY, Jiang JX. Clinical relevance of single nucleotide polymorphisms of the high mobility group box 1 protein gene in patients with major trauma in southwest China. Surgery. 2012 Mar;151(3):427-36. doi: 10.1016/j.surg.2011.07.075. Epub 2011 Nov 1. PMID 22047946
- [Result] Zhang AQ, Zeng L, Gu W, Zhang LY, Zhou J, Jiang DP, Du DY, Hu P, Yang C, Yan J, Wang HY, Jiang JX. Clinical relevance of single nucleotide polymorphisms within the entire NLRP3 gene in patients with major blunt trauma. Crit Care. 2011;15(6):R280. doi: 10.1186/cc10564. Epub 2011 Nov 23. PMID 22112657
- [Result] Zeng L, Gu W, Zhang AQ, Zhang M, Zhang LY, Du DY, Huang SN, Jiang JX. A functional variant of lipopolysaccharide binding protein predisposes to sepsis and organ dysfunction in patients with major trauma. Ann Surg. 2012 Jan;255(1):147-57. doi: 10.1097/SLA.0b013e3182389515. PMID 22167001
- [Result] Zeng L, Zhang AQ, Gu W, Zhou J, Zhang LY, Du DY, Zhang M, Wang HY, Jiang JX. Identification of haplotype tag SNPs within the whole myeloid differentiation 2 gene and their clinical relevance in patients with major trauma. Shock. 2012 Apr;37(4):366-72. doi: 10.1097/SHK.0b013e3182498c8f. PMID 22266968
- [Result] Zhang AQ, Gu W, Zeng L, Zhang LY, Du DY, Zhang M, Hao J, Yue CL, Jiang J. Genetic variants of microRNA sequences and susceptibility to sepsis in patients with major blunt trauma. Ann Surg. 2015 Jan;261(1):189-96. doi: 10.1097/SLA.0000000000000687. PMID 24743625
- [Result] Zeng L, Du J, Gu W, Zhang AQ, Wang HY, Wen DL, Qiu L, Yang XT, Sun JH, Zhang M, Hao J, Jiang JX. Rs1800625 in the receptor for advanced glycation end products gene predisposes to sepsis and multiple organ dysfunction syndrome in patients with major trauma. Crit Care. 2015 Jan 9;19(1):6. doi: 10.1186/s13054-014-0727-2. PMID 25572180
- [Result] Pan W, Zhang AQ, Gu W, Gao JW, Du DY, Zhang LY, Zeng L, Du J, Wang HY, Jiang JX. Identification of haplotype tag single nucleotide polymorphisms within the nuclear factor-kappaB family genes and their clinical relevance in patients with major trauma. Crit Care. 2015 Mar 20;19(1):95. doi: 10.1186/s13054-015-0836-6. PMID 25880845
- [Result] Gao JW, Zeng L, Zhang AQ, Wang X, Pan W, Du DY, Zhang LY, Gu W, Jiang JX. Identification of Haplotype Tag Single-Nucleotide Polymorphisms within the PPAR Family Genes and Their Clinical Relevance in Patients with Major Trauma. Int J Environ Res Public Health. 2016 Mar 26;13(4):374. doi: 10.3390/ijerph13040374. PMID 27023591
- [Result] Zhang H, Lu Y, Sun G, Teng F, Luo N, Jiang J, Wen A. The common promoter polymorphism rs11666254 downregulates FPR2/ALX expression and increases risk of sepsis in patients with severe trauma. Crit Care. 2017 Jul 6;21(1):171. doi: 10.1186/s13054-017-1757-3. PMID 28679406
- [Result] Zhang A, Gu W, Lu H, Zeng L, Zhang L, Du D, Hao J, Wen D, Wang X, Jiang J. Genetic contribution of suppressor of cytokine signalling polymorphisms to the susceptibility to infection after traumatic injury. Clin Exp Immunol. 2018 Oct;194(1):93-102. doi: 10.1111/cei.13160. Epub 2018 Sep 9. PMID 29920655
- [Derived] Wang J, Wen D, Zeng S, Du J, Cui L, Sun J, Chen G, Zeng L, Du D, Zhang L, Deng J, Jiang J, Zhang A. Cytokine Biomarker Phenotype for Early Prediction and Triage of Sepsis in Blunt Trauma Patients. J Surg Res. 2023 Mar;283:824-832. doi: 10.1016/j.jss.2022.10.059. Epub 2022 Dec 5. PMID 36915009
- [Derived] Sun J, Zhang H, Liu D, Cui L, Wang Q, Gan L, Wen D, Wang J, Du J, Huang H, Zhang A, Deng J, Jiang J, Zeng L. A Functional Variant of CXCL16 Is Associated With Predisposition to Sepsis and MODS in Trauma Patients: Genetic Association Studies. Front Genet. 2021 Sep 3;12:720313. doi: 10.3389/fgene.2021.720313. eCollection 2021. PMID 34539750
- [Derived] Lu H, Zhang A, Wen D, Du J, Sun J, Qiao L, Du D, Gu W, Jiang J. Plasma Vanin-1 as a Novel Biomarker of Sepsis for Trauma Patients: A Prospective Multicenter Cohort Study. Infect Dis Ther. 2021 Jun;10(2):739-751. doi: 10.1007/s40121-021-00414-w. Epub 2021 Feb 23. PMID 33624223
- [Derived] Lu H, Wen D, Sun J, Zeng L, Du J, Du D, Zhang L, Deng J, Jiang J, Zhang A. Enhancer polymorphism rs10865710 associated with traumatic sepsis is a regulator of PPARG gene expression. Crit Care. 2019 Dec 30;23(1):430. doi: 10.1186/s13054-019-2707-z. PMID 31888703